CLINICAL TRIAL: NCT06619626
Title: The Effect of Alveolar Recruitment on Perioperative Outcomes in Obese Patients in Major Gynaecological Cancer Surgery: a Prospective Randomised Controlled Trial
Brief Title: Alveolar Recruitment in Obese Patients in Major Gynaecological Cancer Surgery
Status: Recruiting | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Duygu Akyol, Principal Investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: 2023-583
Record Dates: First submitted 2024-09-23; First posted 2024-10-01 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Gynecologic Cancers
Keywords: gynecologic cancer surgery; alveolar recruitment strategy; positive end-expiratory pressure
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1, lung protective ventilation with alveolar recruitment: In mechanical ventilation volume controlled ventilation (VCV) mode, tidal volume (TV) is 6-8 ml/kg according to ideal body weight, positive end expiratory pressure (PEEP): 8 cmH2O, end tidal carbon dioxide pressure (etCO2): 35-45 mmHg, the number of breaths will be adjusted and ventilation will be started. After 10 minutes of ventilation, alveolar recruitment manoeuvre will be started by switching the mechanical ventilator to pressure controlled ventilation (PCV) mode in patients in whom alveolar recruitment strategy (ARS) will be applied. PEEP will be 30 cmHg with 2 unit increases in PEEP for 2 minutes each ventilation will be applied until PEEP reaches 20. When the mean arterial pressure decreases more than 20%, recruitment will be terminated. PEEP will be restored when PEEP 20 is reached. Mechanical ventilation will be switched to VCV mode.
  Interventions: Device: alveolar recruitment strategy applied group; Drug: group without alveolar recruitment strategy
- Group 2, lung protective ventilation without alveolar recruitment: In mechanical ventilation volume controlled ventilation (VCV) mode, tidal volume (TV) is 6-8 ml/kg according to ideal body weight, positive end expiratory pressure (PEEP): 8 cmH2O, end tidal carbon dioxide pressure (etCO2): 35-45 mmHg, ventilation will be provided by adjusting the number of breaths.
  Interventions: Device: alveolar recruitment strategy applied group; Drug: group without alveolar recruitment strategy

INTERVENTIONS:
Device: alveolar recruitment strategy applied group — the effect of alveolar recruitment strategy on the mechanical parameters of the patients
Drug: group without alveolar recruitment strategy — effect on mechanical parameters of patients without alveolar recruitment strategy

SUMMARY:
In this study, the investigators planned to evaluate the effect of alveolar recruitment strategy primarily on postoperative pulmonary complications in obese patients undergoing lung protective ventilation in major open gynaeco-oncological surgeries. Our other aim was to evaluate perioperative haemodynamics, respiratory mechanics,inpatient length of stay.

DETAILED DESCRIPTION:
In the gynaecological oncology clinic of our hospital, open major surgeries for endometrial or ovarian cancer are performed very frequently. In these surgeries, the abdomen is open to the operating theatre environment and the lithotomy and trendelenburg position may have negative consequences on the respiratory system in patients. Intraoperative lung protective ventilation strategies are recommended to reduce postoperative pulmonary complications. In the lung protective ventilation strategy, positive end-expiratory pressure is recommended in addition to 6-8 ml/kg tidal volume according to ideal body weight. In addition, alveolar recruitment strategy can be applied. For this purpose, the investigators planned to evaluate the effect of alveolar recruitment strategy on postoperative pulmonary complications in patients who underwent lung protective ventilation in major open gynaecooncological surgeries. Our secondary aim was to evaluate perioperative haemodynamics, respiratory mechanics, inpatient length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASAII and III
* BMI>30 kg/m2 ,<40 kg/m2
* Patients with an ARISCAT risk score of 26-44

Exclusion Criteria:

* Patients with an Assessment of Respiratory Risk in Surgical Patients in Catalonia (ARISCAT) risk score > 44
* BMI > 40 kg/m2 patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — patients undergoing major gynaecooncological surgery
Study Population: As a result of power analysis, the minimum sample size was determined as 16 for each group with an effect size of 1.2, a 5% margin of error and 95% power. We planned 20 patients for each group due to data losses and deficiencies.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
postoperative pulmonary complications | 24 hours postoperatively
  Our primary aim was to compare the presence of postoperative pulmonary complications. The presence of these pulmonary complications will be compared between preoperative chest X-ray and postoperative day 1 X-ray imaging in patients with Assess Respiratory Risk in Surgical Patients in Catalonia (ARISCAT) risk score below 44.

SECONDARY OUTCOMES:
intraoperative haemodynamic parameters | intraoperatively
  Our secondary aim was to evaluate intraoperative haemodynamic parameter(mean arterial pressure) in alveolar recruitment strategy in lung-protective ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Akyol, Principal Investigator — Başakşehir Çam & Sakura City Hospital
Locations (1):
- Duygu Akyol, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pereira SM, Tucci MR, Morais CCA, Simoes CM, Tonelotto BFF, Pompeo MS, Kay FU, Pelosi P, Vieira JE, Amato MBP. Individual Positive End-expiratory Pressure Settings Optimize Intraoperative Mechanical Ventilation and Reduce Postoperative Atelectasis. Anesthesiology. 2018 Dec;129(6):1070-1081. doi: 10.1097/ALN.0000000000002435. PMID 30260897
- [Background] Park SH. Perioperative lung-protective ventilation strategy reduces postoperative pulmonary complications in patients undergoing thoracic and major abdominal surgery. Korean J Anesthesiol. 2016 Feb;69(1):3-7. doi: 10.4097/kjae.2016.69.1.3. Epub 2016 Jan 28. PMID 26885294
- [Background] Spieth PM, Guldner A, Uhlig C, Bluth T, Kiss T, Conrad C, Bischlager K, Braune A, Huhle R, Insorsi A, Tarantino F, Ball L, Schultz MJ, Abolmaali N, Koch T, Pelosi P, Gama de Abreu M; PROtective Ventilation (PROVE) Network. Variable versus conventional lung protective mechanical ventilation during open abdominal surgery (PROVAR): a randomised controlled trial. Br J Anaesth. 2018 Mar;120(3):581-591. doi: 10.1016/j.bja.2017.11.078. Epub 2017 Dec 1. PMID 29452815